CLINICAL TRIAL: NCT06548607
Title: Clinical Study on Targeted CD19 or CD19-BCMA CAR-T Therapy for Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-04
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: SLE (Systemic Lupus); Systemic Sclerosis; ANCA Associated Vasculitis; Idiopathic Inflammatory Myopathies; Sjogren's Syndrome; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Sjogren's Syndrome; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): RD06-04；RD06-05
  Interventions: Drug: RD06-04 or RD06-05 CART Cell Injection

INTERVENTIONS:
Drug: RD06-04 or RD06-05 CART Cell Injection — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

SUMMARY:
This is an open clinical pharmacological translational Research Study, aiming to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of RD06-04 or RD06-05 in patients with active SLE, SSc, AAV, IIM and pSS.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study and signed the informed consent form.
2. Age ≥18 years old and ≤70 years old, both sexes.
3. Organ function and laboratory tests:

   1. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN), total bilirubin (TBIL) ≤2×ULN (except Gilbert's syndrome).
   2. Renal function: creatinine ≤1.5×ULN or creatinine clearance ≥40 ml/min.
   3. Blood routine: neutrophil count ≥1×109/L, hemoglobin ≥60g/L, platelet count ≥20×109/L, lymphocyte count >0.3×109/L.
   4. Coagulation: international normalized ratio (INR) ≤ 1.5×ULN, or prothrombin time (PT) ≤ 1.5×ULN.
   5. Oxygen saturation (SpO2) ≥92% at rest in room air.
   6. Left ventricular ejection fraction (LVEF) ≥50% on echocardiography.
4. Negative serum or urine pregnancy test results in female subjects of childbearing potential at screening.
5. Women of childbearing potential must agree to use a highly effective method of contraception for at least 28 days before initiation of elution and up to 12 months after RD06-04 reinfusion. Men of childbearing potential had to agree to the use of an effective barrier method of contraception from the initiation of lymphoidectomy until 12 months after reinfusion of RD06-04 and had to refrain from donating semen or sperm throughout the trial.

SLE Patient Inclusion Criteria:

1. A definitive diagnosis of SLE according to the 2019 European League Against Rheumatism (EULAR) / American College of Rheumatology (ACR) classification criteria or the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria.
2. Positive antinuclear antibodies (ANA) at screening, and/or positive anti-double-stranded DNA (anti-dsDNA) antibodies, and/or positive anti-Smith antibodies.
3. A SLEDAI-2K score >6 at screening, and a 'clinical' SLEDAI-2K score ≥4.

SSc Patient Inclusion Criteria:

1. Diagnosed with SSc according to the 2013 ACR/EULAR classification criteria.
2. Diagnosed with diffuse cutaneous SSc at screening, with a disease duration ≤6 years.

AAV Patient Inclusion Criteria:

1. Meeting the diagnostic criteria for ANCA-associated vasculitis established by the 2022 ACR/EULAR, including Microscopic Polyangiitis (MPA), Granulomatosis with Polyangiitis (GPA), and Eosinophilic Granulomatosis with Polyangiitis (EGPA).
2. Positive testing for ANCA-associated antibodies 3 months before screening or at screening (specifically, positive anti-myeloperoxidase antibodies, MPO-ANCA, or positive anti-proteinase 3 antibodies, PR3-ANCA).

IIM Patients Inclusion Criteria:

1. Diagnosed with IIM according to the 2017 ACR/EULAR classification criteria (including probable or definite diagnosis, i.e., probability ≥55%), including subtypes such as Dermatomyositis (DM), Anti-Synthetase Syndrome (ASS), and Immune-Mediated Necrotizing Myopathy (IMNM).
2. Patients in the active phase, defined as those with at least 2 of the following six core set measures being abnormal: decreased muscle strength (MMT-8 <142), Physician Global Assessment (PhGA, 10cm VAS) ≥2cm, Patient Global Assessment (PtGA, 10cm VAS) ≥2cm, Extramuscular Disease Activity Total Score (assessed using the MDAAT scoring tool) ≥2cm, Health Assessment Questionnaire (HAQ) ≥0.25, and Creatine Kinase (CK) muscle enzyme levels ≥1.5×ULN

Sjögren's Syndrome (SS) Patient Inclusion Criteria:

1. Diagnosed with primary Sjögren's Syndrome according to the 2016 ACR/EULAR classification criteria.
2. Positive for anti-SSA/Ro antibodies detected 3 months before screening or at screening.
3. A score of ≥5 on the European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) at screening.

Exclusion Criteria:

1. SLE Patients: Those with uncontrolled lupus crisis within the 8 weeks prior to screening, including rapidly progressive lupus nephritis, severe neuropsychiatric lupus, severe hemolytic anemia, severe immune thrombocytopenia, agranulocytosis, severe cardiac damage, severe lupus pneumonia, severe lupus hepatitis, and severe vasculitis, as assessed by the investigator as unsuitable to participate in this study.
2. IIM Patients: Presence of severe rhabdomyolysis or CK levels ≥120×ULN at screening.
3. Patients with severe asthma or Chronic Obstructive Pulmonary Disease (COPD) are eligible. Patients with mild or moderate asthma or COPD who are receiving stable treatment can also be enrolled.
4. There has been an active infection requiring systemic treatment within 2 weeks prior to the urethral irrigation, such as infectious pneumonia, tuberculosis, etc.
5. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA in peripheral blood; positive for hepatitis C virus (HCV) antibody with detectable HCV RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis antibody.
6. Pregnant or breastfeeding women.
7. Any condition that, in the investigator's opinion, may affect study participation, pose a safety risk to the patient, or potentially confound the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2027-07-29 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (TEAEs), serious adverse events (SAEs), and adverse events of particular concern (AESI) during treatment | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Third the People's Hospital of Bengbu, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No